CLINICAL TRIAL: NCT03612804
Title: Promoting Smoking Cessation in Lung Cancer Screening Through Proactive Treatment
Acronym: PROACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 16-071
Record Dates: First submitted 2018-07-23; First posted 2018-08-02 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Smoking Reduction; Tobacco Use; Tobacco Smoking; Tomography; Lung Diseases; Lung Neoplasms
Keywords: smoking cessation; lung cancer screening; telephone counseling; quitline
MeSH Terms: conditions — Smoking Reduction; Tobacco Use; Tobacco Smoking; Lung Diseases; Lung Neoplasms; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unstructured care (No Intervention): Providers in this arm will continue to provide care as usual during lung cancer screening, with no intervention from the study team.
- Proactive care (Experimental): Providers in this arm will receive guidance from the study team about offering lung cancer screening patients proactive cessation care, including cessation medications and behavioral telephone counseling.
  Interventions: Behavioral: Unsigned note to provider about cessation medication prescription; Behavioral: Proactive Telephone Counseling from VA Quitline

INTERVENTIONS:
Behavioral: Unsigned note to provider about cessation medication prescription — For patients of providers assigned to the proactive study group, a local coordinator will review the patient's cessation medication history. If the patient is not currently being provided cessation support medication, the coordinator will enter a note for the provider about the recommended medication indicated by VA formulary guidelines.
  Arms: Proactive care
Behavioral: Proactive Telephone Counseling from VA Quitline — Patients of providers assigned to the proactive study group will be contacted by specially trained counselors at the VA Quitline. Counselors will attempt to provide two sessions of proactive telephone support.
  Arms: Proactive care

SUMMARY:
This pragmatic trial will evaluate the value of routinely providing proactive smoking cessation support to current smokers as a part of participating in lung cancer screening within Veterans Health Administration.

DETAILED DESCRIPTION:
This trial is a pragmatic randomized trial targeting the care of current smokers who are participating in lung cancer screening at two VA sites. Primary care providers at these sites will be randomized, and half will be offered tools to help integrate proactive smoking cessation support into the lung cancer screening process. Key proactive elements include proactive telephone outreach to all current smokers by a VA Quitline counselor that follows mailed results letters, and providing providers guidance in offering proactive cessation medication support as part of the lung cancer screening process.

ELIGIBILITY:
Inclusion Criteria:

* Providers who schedule patients for a lung cancer screening at either of the two VA sites.
* Patients who participate in lung cancer screening and are current smokers at the time of scheduling their screening exam.

Exclusion Criteria:

* Providers who currently systematically prescribe cessation support medication to all current smokers will be excluded.
* Patients with urgent findings requiring biopsy/immediate attention on the screening CT will be excluded.
* Patients with a prior diagnosis of lung cancer or who are receiving active therapy for any cancer, except skin cancer, will be excluded.
* Patients previously diagnosed with cognitive impairment, dementia, or severe behavioral disorders, or have an indication in chart review of difficulty communicating or participating in telephone counseling sessions will be excluded.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 944 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven B Zeliadt, PhD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (3):
- United States (3):
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The investigators anticipate publishing the findings alongside other similar trials funded by NCI through the Smoking Cessation within the Context of Lung Cancer Screening (SCALE) collaboration, with journals that will likely require concurrent publication of de-identified datasets.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified final datasets will be made available through publisher portals or other repositories identified by SCALE collaboration for ensuring dissemination and publication of trial findings upon completion of the study (2022). Preliminary (de-identified) datasets, study protocol, and statistical analysis plans may be made available to other researchers in the SCALE collaboration throughout the duration of the project.
Access Criteria: Access will only be provided as necessary to allow transparency and evaluation of the results originally obtained by the Principal Investigator who generated the data or to expand upon the work. This assumes the recipient has knowledge, training and resources to adequately design and conduct the studies replicating the original work, or can otherwise determine the validity of results by reviewing the data provided.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a cluster-randomized trial in which providers were randomized to one of two care arms. Patient participants were assigned to an arm based on their provider's care assignment.
Pre-assignment Details: 142 providers and 3,503 patients were screened for eligibility. 26 providers were excluded (19 opt-out before enrolling any patients, 7 not primary care providers) and 2,675 patients were excluded (1,865 not meeting initial inclusion/exclusion criteria, 366 no show to LCS, 178 CT scan not LCS, 130 lung-RADS 4, 87 no copay coverage, 9 provider retired/withdrawn before LCS, 40 no local coordinator to enter notes/COVID complications).
  116 providers and 828 patients were randomized.
Groups:
- Unstructured Care: Providers: Providers in this arm will continue to provide care as usual during lung cancer screening, with no intervention from the study team.
  Patients seen by these providers who receive lung cancer screening will be assigned to the unstructured care arm.
- Unstructured Care: Patients: Providers in this arm will continue to provide care as usual during lung cancer screening, with no intervention from the study team.
- Proactive Care: Providers: Providers in this arm will receive guidance from the study team about offering lung cancer screening patients proactive cessation care, including cessation medications and behavioral telephone counseling.
  Note to provider about cessation medication prescription: For patients of providers assigned to the proactive study group, a local coordinator will review the patient's cessation medication history. If the patient is not currently being provided cessation support medication, the coordinator will enter a note for the provider about the recommended medication indicated by VA formulary guidelines.
  Proactive Telephone Counseling from VA Quitline: Patients of providers assigned to the proactive study group will be contacted by specially trained counselors at the VA Quitline. Counselors will attempt to provide two sessions of proactive telephone support.
  Patients seen by these providers who receive lung cancer screening will be assigned to the proactive care arm.
- Proactive Care: Patients: Providers in this arm will receive guidance from the study team about offering lung cancer screening patients proactive cessation care, including cessation medications and behavioral telephone counseling.
  Note to provider about cessation medication prescription: For patients of providers assigned to the proactive study group, a local coordinator will review the patient's cessation medication history. If the patient is not currently being provided cessation support medication, the coordinator will enter a note for the provider about the recommended medication indicated by VA formulary guidelines.
  Proactive Telephone Counseling from VA Quitline: Patients of providers assigned to the proactive study group will be contacted by specially trained counselors at the VA Quitline. Counselors will attempt to provide two sessions of proactive telephone support.
Period: Overall Study
Arm/Group | Unstructured Care: Providers | Unstructured Care: Patients | Proactive Care: Providers | Proactive Care: Patients
Started | 47 | 422 | 69 | 406
Completed | 46 | 412 | 60 | 378
Not Completed | 1 | 10 | 9 | 28
Not completed — Death | 0 | 7 | 0 | 8
Not completed — Medication copay coverage issues | 0 | 0 | 0 | 17
Not completed — Not current smoker at time of screening | 0 | 1 | 0 | 3
Not completed — Non-veteran status | 0 | 1 | 0 | 0
Not completed — Misassignment to a proactive arm provider | 0 | 1 | 0 | 0
Not completed — Provider retired from VA | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 0
Not completed — Provider involved with study activities | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Proactive Care: Providers: Providers in this arm will receive guidance from the study team about offering lung cancer screening patients proactive cessation care, including cessation medications and behavioral telephone counseling.
  Unsigned note to provider about cessation medication prescription: For patients of providers assigned to the proactive study group, a local coordinator will review the patient's cessation medication history. If the patient is not currently being provided cessation support medication, the coordinator will enter a note and unsigned order for the provider about the recommended medication indicated by VA formulary guidelines.
  Proactive Telephone Counseling from VA Quitline: Patients of providers assigned to the proactive study group will be contacted by specially trained counselors at the VA Quitline. Counselors will attempt to provide two sessions of proactive telephone support.
  Patients seen by these providers who receive lung cancer screening will be assigned to the proactive care arm.
- Proactive Care: Patients: Providers in this arm will receive guidance from the study team about offering lung cancer screening patients proactive cessation care, including cessation medications and behavioral telephone counseling.
  Unsigned note to provider about cessation medication prescription: For patients of providers assigned to the proactive study group, a local coordinator will review the patient's cessation medication history. If the patient is not currently being provided cessation support medication, the coordinator will enter a note and unsigned order for the provider about the recommended medication indicated by VA formulary guidelines.
  Proactive Telephone Counseling from VA Quitline: Patients of providers assigned to the proactive study group will be contacted by specially trained counselors at the VA Quitline. Counselors will attempt to provide two sessions of proactive telephone support.
- Total: Total of all reporting groups
Arm/Group | Unstructured Care: Providers | Unstructured Care: Patients | Proactive Care: Providers | Proactive Care: Patients | Total
Number analyzed (Participants) | 47 | 412 | 69 | 378 | 906
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data not collected for providers.
  years
    number analyzed (Participants) | 0 | 412 | 0 | 378 | 790
    (all) |  | 66.7 (5.9) |  | 66.6 (6.5) | 66.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not collected for providers.
  Participants
    number analyzed (Participants) | 0 | 412 | 0 | 378 | 790
    Female |  | 19 |  | 18 | 37
    Male |  | 393 |  | 360 | 753
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected for providers.
  Participants
    number analyzed (Participants) | 0 | 412 | 0 | 378 | 790
    Hispanic or Latino |  | 20 |  | 36 | 56
    Not Hispanic or Latino |  | 382 |  | 336 | 718
    Unknown or Not Reported |  | 10 |  | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected for providers.
  Participants
    number analyzed (Participants) | 0 | 412 | 0 | 378 | 790
    American Indian or Alaska Native |  | 1 |  | 3 | 4
    Asian |  | 2 |  | 4 | 6
    Native Hawaiian or Other Pacific Islander |  | 1 |  | 1 | 2
    Black or African American |  | 50 |  | 104 | 154
    White |  | 346 |  | 246 | 592
    More than one race |  | 2 |  | 5 | 7
    Unknown or Not Reported |  | 10 |  | 15 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 412 | 69 | 378 | 906

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Smoking Abstinence
Description: The primary outcome measure is self-reported abstinence from smoking 12 months after lung cancer screening, using information obtained from study surveys and electronic medical records. This measure only applies to patient enrollees.
Time Frame: 12 months after lung cancer screening visit
Population: Enrolled participants with complete outcome data. The overall number of participants analyzed is lower than enrolled participants due to missing survey/electronic medical records data.
Measure: Count of Participants; unit: Participants
Groups:
- Proactive Care: Patients: Providers in this arm will receive guidance from the study team about offering lung cancer screening patients proactive cessation care, including cessation medications and behavioral telephone counseling.
  Unsigned note to provider about cessation medication prescription: For patients of providers assigned to the proactive study group, a local coordinator will review the patient's cessation medication history. If the patient is not currently being provided cessation support medication, the coordinator will enter a note for the provider about the recommended medication indicated by VA formulary guidelines.
  Proactive Telephone Counseling from VA Quitline: Patients of providers assigned to the proactive study group will be contacted by specially trained counselors at the VA Quitline. Counselors will attempt to provide two sessions of proactive telephone support.
Arm/Group | Unstructured Care: Patients | Proactive Care: Patients
Number analyzed (Participants) | 359 | 322
Participants | 50 | 51
Statistical Analysis 1: Comparison: Unstructured Care: Patients vs Proactive Care: Patients; Test type: Superiority; p = 0.83, Regression, Logistic — P-value not adjusted for multiple comparisons. A priori threshold for statistical significance was 0.05; Logistic regression model with random intercept for provider and main effect term for study site; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.67 to 1.64] — Proactive care arm represents numerator of odds ratio, unstructured care arm represents denominator of odds ratio

2. Secondary Outcome: Cost of Smoking Cessation Care
Description: Costs of implementing smoking cessation care from lung cancer screening to 12 months post-lung cancer screening will be monitored in both the unstructured and proactive care arms. Cost of implementing smoking cessation care is defined as the sum of the cost of behavioral counseling, cost of pharmacotherapies, and cost of intervention staff effort. This measure only applies to patient enrollees.
Time Frame: Time period from lung cancer screening through 12 months after lung cancer screening
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Unstructured Care: Patients | Proactive Care: Patients
Number analyzed (Participants) | 412 | 378
dollars | 34.1 (159.1) | 384.2 (161.1)

3. Secondary Outcome: Patients' Experience With Telephone Counseling
Description: Binary variable for whether participant reported being either very satisfied or somewhat satisfied with VA Quitline telephone counseling. This measure only applies to patient enrollees in the proactive arm.
Time Frame: 3 months after lung cancer screening visit
Population: Subset of participants in the Proactive Care arm who responded to the 3 month survey and rated their satisfaction with VA Quitline telephone counseling.
Measure: Count of Participants; unit: Participants
Arm/Group | Proactive Care: Patients
Number analyzed (Participants) | 98
Participants | 34

4. Secondary Outcome: Patients' Motivational Assessment
Description: Surveys will assess patient motivation to quit smoking on a scale from 0-10 (higher scores indicate higher motivation to quit smoking). This measure only applies to patient enrollees.
Time Frame: 3 months after lung cancer screening visit
Population: Subset of overall sample who responded to the 3 month survey and rated their motivation to quit smoking.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unstructured Care: Patients | Proactive Care: Patients
Number analyzed (Participants) | 106 | 97
score on a scale | 7.54 (3.01) | 7.95 (3.05)

5. Secondary Outcome: Patients' Perception of Susceptibility to Harm
Description: Surveys will assess patients' perceived susceptibility to the harmful effects of smoking and perception of screening as protective. Patients were asked 5 questions related to smoking and screening, and an overall score based on the sum of correct answers was calculated. Scores range from 0-5 (higher scores indicate greater knowledge about harmful effects of smoking and benefits of screening). This measure only applies to patient enrollees.
Time Frame: 3 months after lung cancer screening visit
Population: Subset of overall sample who responded to the 3 month survey and rated their perceived susceptibility to the harmful effects of smoking and perception of screening as protective.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unstructured Care: Patients | Proactive Care: Patients
Number analyzed (Participants) | 103 | 91
score on a scale | 1.97 (1.11) | 2.09 (1.02)

6. Secondary Outcome: Patients' Self-efficacy Assessment
Description: Surveys will assess patients' self-efficacy for quitting smoking on a scale from 0-10 (higher scores indicate greater self-efficacy for quitting smoking). This measure only applies to patient enrollees.
Time Frame: 3 months after lung cancer screening visit
Population: Subset of overall sample who responded to the 3 month survey and rated their self-efficacy for quitting smoking.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unstructured Care: Patients | Proactive Care: Patients
Number analyzed (Participants) | 100 | 92
score on a scale | 5.7 (3.3) | 6.5 (3.1)

7. Secondary Outcome: Patients' Motivational Assessment
Description: as for outcome 4
Time Frame: 12 months after lung cancer screening visit
Population: Subset of overall sample who responded to the 12 month survey and rated their motivation to quit smoking.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unstructured Care: Patients | Proactive Care: Patients
Number analyzed (Participants) | 116 | 113
score on a scale | 7.48 (2.95) | 7.3 (3.2)

8. Secondary Outcome: Patients' Self-efficacy Assessment
Description: as for outcome 6
Time Frame: 12 months after lung cancer screening visit
Population: Subset of overall sample who responded to the 12 month survey and rated their self-efficacy for quitting smoking.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Unstructured Care: Patients | Proactive Care: Patients
Number analyzed (Participants) | 117 | 114
score on a scale | 5.8 (3.4) | 6.1 (3.3)

ADVERSE EVENTS:
Time Frame: 1 year following LCS date
Description: All-cause mortality during the 1 year period following LCS was assessed for all patients (providers not assessed). Serious and other non-serious adverse events were not assessed.
Groups:
- Proactive Care: Providers: Providers in this arm will receive guidance from the study team about offering lung cancer screening patients proactive cessation care, including cessation medications and behavioral telephone counseling.
  Unsigned note to provider about cessation medication prescription: For patients of providers assigned to the proactive study group, a local coordinator will review the patient's cessation medication history. If the patient is not currently being provided cessation support medication, the coordinator will enter a note for the provider about the recommended medication indicated by VA formulary guidelines.
  Proactive Telephone Counseling from VA Quitline: Patients of providers assigned to the proactive study group will be contacted by specially trained counselors at the VA Quitline. Counselors will attempt to provide two sessions of proactive telephone support.
  Patients seen by these providers who receive lung cancer screening will be assigned to the proactive care arm.
Arm/Group | Unstructured Care: Providers | Unstructured Care: Patients | Proactive Care: Providers | Proactive Care: Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 7/422 | 0/0 | 8/406
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We originally planned to base our smoking cessation outcome on biochemically-confirmed 7-day smoking abstinence. Due to the COVID-19 pandemic, it was not possible to perform the saliva cotinine testing needed for biochemically confirmed abstinence, and no biochemical data were collected. Instead, we updated our study protocol to use a combination of survey and electronic medical record data to determine smoking status at 12 months post-lung cancer screening as our primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT03612804/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03612804/SAP_001.pdf